CLINICAL TRIAL: NCT03853993
Title: Open Phase I and Randomized, Double-blind, Controlled Phase III Clinical Trial to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine in Healthy Subjects Aged Over 3 Years.
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine (15µg/0.5ml)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-QINF-3001
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Seasonal Influenza
Keywords: Influenza Vaccine; Quadrivalent; Trivalent
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: The phase I clinical trial has single arm, and the phase III clinical trial has 3 parallel arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group-phase I (Experimental): Quadrivalent influenza vaccine
  Interventions: Biological: Quadrivalent influenza vaccine
- Experimental group-phase III (Experimental): Quadrivalent influenza vaccine
  Interventions: Biological: Quadrivalent influenza vaccine
- Control group-1-phase III (Active Comparator): Trivalent influenza vaccine (contains B/Victoria strain)
  Interventions: Biological: Trivalent influenza vaccine (contains B/Victoria strain)
- Control group-2-phase III (Active Comparator): Trivalent influenza vaccine (contains B/Yamagata strain)
  Interventions: Biological: Trivalent influenza vaccine (contains B/Yamagata strain)

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — Received single dose QIV (15µg/0.5ml)
  Arms: Experimental group-phase I; Experimental group-phase III
Biological: Trivalent influenza vaccine (contains B/Victoria strain) — Received single dose TIV which contains B/Victoria strain (15µg/0.5ml)
  Arms: Control group-1-phase III
Biological: Trivalent influenza vaccine (contains B/Yamagata strain) — Received single dose TIV which contains B/Yamagata strain (15µg/0.5ml)
  Arms: Control group-2-phase III

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of quadrivalent influenza vaccine in healthy subjects aged over 3 years

DETAILED DESCRIPTION:
This study is a phase I& III clinical trial. Phase I is open-labelled, and phase III is randomized, double-blind, active-controlled. The purpose of this study is to evaluate the safety and immunogenicity of the quadrivalent influenza vaccine (QIV) (experimental vaccine) manufactured by Sinovac Biotech Co., Ltd in subjects aged over 3 years. In phase I, 60 volunteers received single dose QIV (15µg/0.5ml). In phase III, 2320 volunteers were assigned to receive single dose QIV (15µg/0.5ml) or two commercial trivalent influenza vaccines (TIVs) (15µg/0.5ml) in a ratio of 2:1:1. The commercial TIVs were also manufactured by Sinovac Biotech Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged ≥3 years;
* Proven legal identity;
* Participants or (and) guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment;

Exclusion Criteria:

* Prior vaccination with influenza vaccine of the current year;
* History of influenza within 6 months prior to study entry;
* Axillary temperature > 37.0 °C;
* History of allergy to any vaccine, or any ingredient of the experimental vaccine, especially eggs, egg albumin, etc.;
* Serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc.;
* Severe/uncontrollable nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* Autoimmune disease or immunodeficiency/immunosuppressive, or any immunosuppressant receipt within 6 months prior to the study entry;
* History of asthma, thyroidectomy, angioedema, diabetes or malignancy;
* No spleen, or functional no spleen, or splenectomy.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2380 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
The lower limit of 95% confidence intervals (95%CI) of the ratio of geometric mean titer of hemagglutination inhibition (HI) antibody titer (experimental group/control group)≥2/3. | 28 days after the injection
  Immunogenicity index, One of the standard to evaluate the experimental vaccine is non-inferior to the control vaccines
The lower limit of 95% CI of the difference of HI antibody seroconversion rate (experimental group-control group)≥-10% | 28 days after the injection
  Immunogenicity index, Another standard to evaluate the experimental vaccine is non-inferior to the control vaccines

SECONDARY OUTCOMES:
The lower limit of 95%CI of the ratio of GMT(experimental group/control group)>1.5 . | 28 days after the injection
  Immunogenicity index, One of the standard to evaluate the experimental vaccine is superior to the control vaccines for specific antigen type
The lower limit of 95% CI of the difference of HI antibody seroconversion rate (experimental group-control group)>10% | 28 days after the injection
  Immunogenicity index, Another standard to evaluate the experimental vaccine is superior to the control vaccines for specific antigen type
The 95% CI lower limit of seroconversion rate of HI antibodies in the subjects aged 3-59 years≥40% | 28 days after the injection
  Immunogenicity index
The 95% CI lower limit of seroconversion rate of HI antibodies in the subjects aged over 60 years≥30% | 28 days after the injection
  Immunogenicity index
The seroprotective rate (HI antibody titer≥1:40) in the subjects aged 3-59 years ≥70% | 28 days after the injection
  Immunogenicity index
The seroprotective rate (HI antibody titer≥1:40) in the subjects aged over 60 years ≥60% | 28 days after the injection
  Immunogenicity index
The geometric mean increase (GMI) in the subjects aged 3-59 years >2.5 | 28 days after the injection
  Immunogenicity index
The geometric mean increase (GMI) in the subjects aged over 60 years >2.0 | 28 days after the injection
  Immunogenicity index
The lower limit of 95%CI of the ratio of GMT(experimental group/control group)≥2/3, in the subjects whose pre-immune HI antibody titer<1:40 | 28 days after the injection
  Immunogenicity index
The lower limit of 95% CI of the difference of HI antibody seroconversion rate (experimental group-control group)≥-10%, in the subjects whose pre-immune HI antibody titer<1:40 | 28 days after the injection
  Immunogenicity index
The incidence of the solicited local and general adverse reactions on day 0-7 | 0-7 days after the injection
  Safety index, The adverse reactions refers to the adverse events which considered related to the vaccination
The incidence of the unsolicited adverse events on day 0-28 | 0-28 days after the injection
  Safety Index
The incidence of the serious adverse events within 6 months after the injection | Within 6 months after the injection
  Safety Index

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Province Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Guanyun Center for Disease Control and Prevention, Lianyungang, Jiangsu
  - Pizhou Center for Disease Control and Prevention, Pizhou, Jiangsu

REFERENCES:
- [Derived] Chu K, Xu K, Tang R, Tian X, Hu J, Yang T, Li C, Hu Y, Zeng G. Immunogenicity and safety of an inactivated quadrivalent influenza vaccine: A randomized, double-blind, controlled phase III study in healthy population aged >/=3 years. Vaccine. 2020 Aug 18;38(37):5940-5946. doi: 10.1016/j.vaccine.2020.06.071. Epub 2020 Jul 27. PMID 32732142